CLINICAL TRIAL: NCT07152158
Title: Effect of Multicomponent Training Combined With Multi-professional Intervention on Health Status in Hypertensive and Normotensive Older Women
Brief Title: Multicomponent Training Combined With Multi-professional Intervention Health Status in Hypertensive and Normotensive Older Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica del Maule (Other)
Collaborators: University of Talca (Other); Universidad de Los Lagos (Other)
Responsible Party: Principal Investigator, Pablo Valdés-Badilla, Principal Investigator, Universidad Católica del Maule
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3.373.307
Record Dates: First submitted 2025-08-22; First posted 2025-09-03 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Older People
Keywords: Biomarkers; Cardiovascular System; Body Composition; Physical Functional Performance

STUDY DESIGN:
Intervention Model Description: The design of this study is descriptive, longitudinal and quasi-experimental in four time points (T0: baseline, T1: 12 weeks, T2: 24 weeks, and T3: 36 weeks) with a frequency of three sessions per week (Monday, Wednesday, and Friday) lasting 60 minutes, which consisted of interventions through MCT, nutritional education, and psychoeducation. The present study was publicized through various communication channels (e.g., television, radio, social media) to recruit participants. Body composition (BFP and FFM), blood pressure (SBP and DBP), biochemical variables (glucose, cholesterol, triglycerides), and physical performance (MIHS, arm curl, 30-second chair stand, 6MWT, and TUG) were evaluated. All measurements were taken in the morning, between 9:00 and 11:00 a.m., and in the same place: Interdisciplinary Laboratory for Health Promotion Interventions (LIIPS) at Cesumar University, Maringa, Paraná Brazil.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- multicomponent training combined (Experimental): The intervention activities consisted of two weekly MCT sessions and one session divided into nutritional and psychological education. The MCT intervention sessions lasted approximately 60 minutes and were conducted on the university premises. The exercises were designed to improve flexibility, strength, mobility, motor coordination, balance, and cardiorespiratory fitness. It should be noted that the MCT program was implemented alternately in indoor and outdoor settings, i.e., one day of the week was devoted to indoor training (gym setting), while another day was devoted to outdoor training (open space).
  Interventions: Other: multicomponent training combined with multi-professional intervention

INTERVENTIONS:
Other: multicomponent training combined with multi-professional intervention — The MCT protocol consisted of an initial three-week period of neuromotor adaptation characterized by low volume and intensity. In the subsequent weeks, a gradual progression of volume and intensity was implemented (Table 1), following a classic linear periodization model (Fleck & Kraemer, 2017; Prestes et al., 2016).

SUMMARY:
Objective: The objective of this study was to analyze the effects of multicomponent training (MCT) combined with multidisciplinary intervention (nutritional and psychoeducation) on body composition, biochemical markers, and physical performance in hypertensive and normotensive older women. Methods: This longitudinal study included 40 hypertensive and normotensive older women. These older women performed MCT for 36 weeks, during which parameters associated with health status were evaluated (body composition: body fat, fat-free mass; cardiovascular variables: systolic blood pressure (SPBP), diastolic blood pressure (DBP); biochemical markers: glucose, LDL-cholesterol, HDL-cholesterol, total cholesterol, triglycerides; physical performance: arm curl, maximal isometric handgrip strength (MIHS), 30-second chair stand, 6-meter walking test (6MWT), and Timed Up and Go (TUG)). at four time points: baseline (T0), 12 weeks (T1), 24 weeks (T2), and 36 weeks (T3). A two-way mixed analysis of variance with repeated measures was performed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older and medical clearance to engage in physical exercise
* Those who demonstrated the capacity to comprehend and carry out instructions in a contextualized way through basic directives;
* Those who were independent, as indicated by a score of at least 43 points on the Chilean Ministry of Health's Preventive Medicine Exam for the Older People
* Those who were able to meet the intervention's attendance requirement of at least 85%.

Exclusion Criteria:

* Diagnosed with debilitating neurological disorders (e.g., Alzheimer's disease or Parkinson's disease)
* Older people with contraindications to physical exercise, and those with cardiac arrhythmias.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 63 (Actual)
Dates: Start 2025-09-17 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Biomarkers analyses | 36 weeks
  The blood collection procedures followed the guidelines of the Clinical Laboratory Standards Institute . The participants were previously instructed to prepare accordingly for the collections which were conducted at the Clinical Analysis Laboratory of the Institution's facilities. After the blood was drawn, they were advised to apply pressure to the puncture site to prevent bruising. The blood samples were distributed into the following tubes: Vacuplast® collection tubes, tubes containing the anticoagulant ethylenediaminetetraacetic acid (EDTA) K2, and tubes with fluoride/EDTA anticoagulant.
Anthropometry | 36 weeks
  The standing height of the participants was measured via a stadiometer (Welmy R - 110®, Santa Bárbara D'Oeste, São Paulo, Brazil) attached to a scale with a maximum capacity of 2.2 meters and an accuracy of 0.1 cm.
Physical performance TUG | 36 weeks
  Following earlier suggestions, the TUG test was conducted. The person must get out of an arm-supported chair, cross a three-meter aisle, turn around, and return to the chair. They must perform three trials and record the best one in seconds. A pair of evaluators measured the time using single-beam photocells (Brower Timing System, Draper, UT, USA), and the best of three trials was utilized for statistical analysis
30-second chair stand | 36 weeks
  Three repetitions were evaluated to retrieve the best performance executed on the 30-chair stand test. Its purpose was to evaluate the lower limbs' muscle strength, and it is executed while seated in a chair, with the arms resting across the chest, for 30 s.
Arm curl Test | 36 weeks
  In the arm-curl test, participants sat on a chair and were asked to flex the elbow of their stronger arm as many times as possible in 30 seconds while holding a 1-kg dumbbell. Participants were instructed to maintain a normal breathing pattern and keep their elbow at their side during the entire test. A single repetition consisted of full elbow flexion from maximal extension
MIHS | 36 weeks
  Previous studies have recommended the use of MIHS testing. The most suitable testing position was determined to be seated, with the forearm and wrist maintained in a neutral position, the elbow flexed at 90◦ and kept close to the torso, the spine properly aligned, and the shoulder relaxed in a neutral position. A handheld dynamometer (Jamar®, PLUS+, Sammons Preston, Patterson Medical, Warrenville, IL, USA) was used to perform the measurements. To accommodate varying hand sizes and ensure effective engagement of the metacarpophalangeal and interphalangeal joints, the dynamometer was set to the first position, allowing contact between the thumb and the proximal phalanx of the index finger. Participants were given a 120 s rest period between each of the three repetitions per hand.
6MWT | 36 weeks
  Heart rate (HR) was recorded at rest and at the end of each minute during the 6MWT using a lightweight telemetric HR monitor. Oxygen saturation (SpO2) was recorded before and after completing the 6MWT using an oximeter and a finger sensor. At the end of the test, distance was measured and, where appropriate, leg fatigue was assessed using a modified Borg scale from 0 to 10.
body composition | 36 weeks
  Body composition was assessed via a tetrapolar bioelectrical impedance analyzer (InBody 570®, Bio space Co. Ltd., Seoul, South Korea), with a capacity of 250 kg and an accuracy of 100 g, following the manufacturer's instructions and establishing recommendations to increase precision and reliability. The following variables were assessed: body weight (kg), BFP, FFM (kg), and body mass index (BMI, kg/m²).

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica del Maule, Talca, Talca, Chile

IPD SHARING:
Plan to Share IPD: No
They will not be shared, since the data will be private only for the researchers, after prior agreement with the ethics committee.